CLINICAL TRIAL: NCT01184729
Title: 6 Minute Propulsion Test Sensitivity to Increased Aerobic Capacity
Status: Completed | Type: Observational
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Mark S. Nash, Ph.D., FACSM, Professor, University of Miami
Other Study IDs: TMP MN 002
Record Dates: First submitted 2010-08-18; First posted 2010-08-19 (Estimated); Last update posted 2014-07-22 (Estimated); Status verified 2014-07

CONDITIONS: Spinal Cord Injury
Keywords: aerobic capacity
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Spinal Cord Injury

SUMMARY:
The goals of this project are to 1)determine the responsiveness of the 6 Minute Push Test (6MPT) and 2) explore the relationship between 6MPT distance and measures of handicap, wheelchair satisfaction, depression, and self-reported avoidance of environmental features.

DETAILED DESCRIPTION:
The 6 minute walk test is a widely used assessment of aerobic capacity, function, and functional change in the ambulatory population. A similar clinical and research outcome instrument that is responsive to changes in aerobic capacity and function are lacking for persons with spinal cord injury (SCI). A 6 minute push test, adapted from the 6 minute walk test may fill the void. The primary aim of this project is to assess if distance traveled in 6 minutes of wheelchair propulsion changes after an increase in aerobic capacity. We hypothesize that participants will push farther in 6 minutes after their aerobic capacity increases. The secondary aim is to explore the correlation between 6MPT distance and handicap, depression, wheelchair satisfaction, and self-reported avoidance of environmental features. We hypothesize increasing 6MPTdistance will be correlated with decreasing depression, decreasing handicap, decreasing self-reported avoidance of environmental features, and increasing wheelchair satisfaction. This is a low risk, high benefit study.

ELIGIBILITY:
Inclusion Criteria:

* T1 or lower injury
* at least 1 year post-injury
* able to self-propel a manual wheelchair
* enrolled in TMP-MN-006

Exclusion Criteria:

* Not enrolled in the IRB approval parent study, "Exercise Treatment of Obesity-Related Secondary Conditions in Adults with Paraplegia", TMP-MN-006
* Unstable angina or myocardial infarction within the past month
* Resting heart rate >120
* Systolic blood pressure > 180 mm Hg
* Diastolic blood pressure > 100 mm Hg

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Community sample of persons with spinal cord injury
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2008-11; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Change in Oxygen uptake during 6 min Push Test From baseline. | Visits 1-4
  Subjects will be prepared by putting a flexible mask over the mouth and nose. Heart rate during testing will be monitored by either three electrodes on the chest or by a monitor strapped around the chest. Heart rate and oxygen consumption during each 6MPT will be measured. Participants will be instructed to propel as far as possible on a 30m loop marked at 3m intervals, with 15m between pylons, and two 180 degree turns. Distance traveled in 6 minutes (m) will be computed by multiplying the number of full laps completed by 15m and adding the distance traveled in the last lap.

CONTACTS AND LOCATIONS:
Overall Officials: Mark S Nash, PhD, Principal Investigator — University of Miami, The Miami Project to Cure Paralysis
Locations (1):
- The Miami Project to Cure Paralysis, Miami, Florida, United States